CLINICAL TRIAL: NCT06173167
Title: Clinical Evaluation of Full Contour Zirconia Chairside CAD/CAM Crowns
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ivoclar Vivadent AG (Industry)
Collaborators: University of Michigan (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: OTCS11686932; HUM00241710 (Other: University of Michigan)
Record Dates: First submitted 2023-12-07; First posted 2023-12-15 (Actual); Last update posted 2024-03-28 (Actual); Status verified 2023-12

CONDITIONS: Dental Disorders Hard Tissues of Teeth; Dental Diseases
Keywords: Dental Caries, Caries
MeSH Terms: conditions — Stomatognathic Diseases; Dental Caries

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- SpeedCEM Plus luted crowns (Experimental): crowns delivered with a self-adhesive, self-curing resin cement (SpeedCEM Plus\Ivoclar Vivadent AG)
  Interventions: Device: Crowns self-adhesively luted
- ZirCAD Cement cemented crowns (Experimental): crowns delivered with a resin modified glass ionomer cement (ZirCAD Cement\Ivoclar Vivadent AG)
  Interventions: Device: Crowns conventionally cemented

INTERVENTIONS:
Device: Crowns self-adhesively luted — After cavity preparation, the zirconia chairside crown will be placed using SpeedCEM Plus. The excess will be light cured with Bluephase G4 in PreCure mode (950 mW/cm^2). After removal of the excess, the luting material margins will be light-cured again for 20s (1200 mW/cm^2).
  Arms: SpeedCEM Plus luted crowns
Device: Crowns conventionally cemented — After cavity preparation, the zirconia chairside crown will be placed using ZirCAD Cement. The excess cement will be removed in the gel phase, either following light curing (5 - 10 seconds per segment) or following self-curing (approximately 2 min after placement). The restoration will be held in position during final curing that is complete 4 min 30 s after placement.
  Arms: ZirCAD Cement cemented crowns

SUMMARY:
This investigation will be a randomized, prospective, longitudinal clinical trial to study the clinical performance of a new monolithic, zirconia material with shade, translucency and material graduation for chairside CAD/CAM crowns. The restorations will be luted either with a self-adhesive luting material or a conventional cement. The crowns will be evaluated for a period of two years.

ELIGIBILITY:
Inclusion Criteria:

* at least 18 years of age
* at least one carious lesion, defective restoration, or fractured portion of the tooth to be restored on a maxillary or mandibular premolar or molar tooth - Each lesion, fracture, or defective restoration should exhibit sufficient size or loss of tooth structure requiring a full crown restoration.
* tooth should have at least one opposing tooth in occlusion and one adjacent tooth with an intact proximal contact
* No more than ten teeth that are endodontically treated may be included in the study, equally divided between the two groups of crowns. All remaining teeth in the study will test vital and be asymptomatic at the beginning of treatment.
* No more than two restorations will be placed per patient

Exclusion Criteria:

* Sensitive teeth
* Teeth with a history of direct or indirect pulp capping procedures
* Patients with significant untreated dental disease to include periodontitis and/or rampant caries
* Women who self-report that they are possibly pregnant, pregnant, or lactating, as elective dental treatment is not indicated at these times
* Patients with a self-reported history of allergies to the materials to be used in the study including composite resin cements or zirconia restorative materials
* Patients unable to return for the recall appointments

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2024-01-08 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Short-term Post-operative Sensitivity | 4 weeks
  assessed by patient's weekly feedback for 4 weeks after the treatment rating sensitivity from 1 "no sensitivity" to 4 "severe discomfort noted routinely with cold or pressure stimulation"

SECONDARY OUTCOMES:
Quality Criteria (modified FDI criteria) | 1 year to 2 years
  assessed following the FDI criteria on a scale from 1 "very good" to 5 "unacceptable" (e.g. post-operative hypersensitivity, surface lustre, Staining, fracture of material, retension, occlusal contour and wear, and colour match of restorations)

CONTACTS AND LOCATIONS:
Overall Officials: Dennis J. Fasbinder, DDS, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan School of Dentistry, Ann Arbor, Michigan, United States